CLINICAL TRIAL: NCT07225205
Title: Home Intravenous Fluid Infusion After Undergoing Radical Cystectomy: A Randomized Controlled Trial
Brief Title: Home Intravenous Fluid Infusion After Undergoing Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00516342
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer; Muscle Invasive Bladder Cancer (MIBC); Muscle Invasive Bladder Cancer Urothelial Carcinoma; Cystectomy
Keywords: Cystectomy; Bladder Cancer; Muscle Invasive Bladder Cancer (MIBC); Fluids; IVF; ERAS
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home IVF + ERAS (Experimental): Patients assigned to the home IVF arm will undergo the investigator's current ERAS pathway, which involves establishing vascular access that can be used for 4 weeks at home. Many patients have existing vascular access via a port which the participant receives for neoadjuvant chemotherapy. If the patient does not have existing access, the JHH Vascular Access Team (VAT) is engaged during the post-operative hospitalization to place a midline catheter, which is a type of peripheral vascular access that is adequate for 4 week durations and is less invasive than central catheters. Once the patient has vascular access, the home care coordinator and social worker are engaged to organize home nursing for wound care, ostomy teaching, and home IVF. At home, the patient receives a 1L bolus of either lactated ringers or normal saline three times a week for four weeks with the participant's home nurse.
  Interventions: Other: Intravenous fluids; Other: ERAS
- ERAS Alone (No Intervention): Patients assigned to not receive home IVF will receive everything in the investigator's current ERAS protocol except the home intravenous fluid program. Patients without preexisting vascular access will not receive a midline catheter post-operatively, however the participant will still receive home care for skilled nursing who will provide wound care, ostomy teaching, and education about perioperative fluid management.

INTERVENTIONS:
Other: Intravenous fluids — At home, the patient receives a 1L bolus of either lactated ringers or normal saline three times a week for four weeks with the patient's home nurse.
  Arms: Home IVF + ERAS
Other: ERAS — Patients assigned to not receive home IVF will receive everything in the investigator's current ERAS protocol except the home intravenous fluid program. Patients without preexisting vascular access will not receive a midline catheter post-operatively, however the participant will still receive home care for skilled nursing who will provide wound care, ostomy teaching, and education about perioperative fluid management.
  Arms: Home IVF + ERAS

SUMMARY:
Radical cystectomy is the standard of care for muscle invasive bladder cancer, however despite advances, it is still associated with high morbidity. Many complications may be driven by dehydration and it is unclear if a home intravenous fluid (IVF) infusion program post-operatively, which is an accepted standard practice, is beneficial. This study is a single institution randomized controlled trial where patients who choose to undergo radical cystectomy for bladder cancer will be randomized to an Enhanced Recovery After Surgery (ERAS) protocol with a home IVF program, consisting of 1 liter (L) of crystalloid fluid three times per week for four weeks, or ERAS protocol alone. The primary outcome will be 90-day hospital re-admissions, with secondary outcomes including 30 and 90 day complications.

DETAILED DESCRIPTION:
The standard of care for patients with muscle-invasive bladder cancer is to undergo a radical cystectomy (RC), bilateral pelvic lymph node dissection and urinary diversion, but this surgery is associated with substantial perioperative morbidity frequently exceeding 60% 90-day complication rates. ERAS protocols have been widely adopted to improve perioperative outcomes in RC. These multimodal pathways reduce length of stay, expedite bowel recovery, and decrease overall complication rates, but have not consistently reduced readmission rates. The most common causes of readmission include dehydration, urinary tract infection, and ileus, with dehydration being a particularly modifiable risk factor.

The ERAS pathway employed at Johns Hopkins Hospital (JHH) utilizes IVF infusion programs to promote hydration in the post-operative period. This is based on both substantial clinical experience that suggest the driver of many hospital re-admissions may be dehydration and a prospective study that found a substantial decrease in 90-day readmission rates with the addition of a home IVF program to the ERAS protocol. However, there is still a paucity of high quality evidence on the addition of a home IVF program to ERAS protocols and this addition is not without its risks, particularly related to the necessity of indwelling venous catheters. Additionally, ERAS protocols for RC were originally developed and validated in the context of open surgical approaches, which are associated with higher intraoperative blood loss and fluid shifts. However, the adoption of robot-assisted RC has led to significantly lower estimated blood loss and reduced transfusion requirements compared to open RC. These improvements in surgical technique may reduce the need for aggressive perioperative fluid replacements. Taken together, this evidence underscores the need for randomized trial evidence to evaluate home IVF programs in RC ERAS protocols.

The study will be a single-blinded prospective randomized controlled trial in patients undergoing RC for bladder cancer. Patients will be randomized in a 1:1 fashion to either receive home IVF or standard peri-operative education related to hydration. This randomization will be stratified based on the urinary diversion the patient receives, which will either be an ileal conduit or a neobladder, and the patient's sex. Patients will be consented pre-operatively by a physician on the research team. The surgeon and surgical team will be blinded to the group assignment before and during the surgery.

Patients assigned to the home IVF arm will undergo the investigator's current ERAS pathway, which involves establishing vascular access that can be used for 4 weeks at home. Many patients have existing vascular access via a port which the participant receives for neoadjuvant chemotherapy. If the patient does not have existing access, the JHH Vascular Access Team (VAT) is engaged during the post-operative hospitalization to place a midline catheter, which is a type of peripheral vascular access that is adequate for 4 week durations and is less invasive than central catheters. Once the patient has vascular access, the home care coordinator and social worker are engaged to organize home nursing for wound care, ostomy teaching, and home IVF. At home, the patient receives a 1L bolus of either lactated ringers or normal saline three times a week for four weeks with the patient's home nurse.

Patients assigned to not receive home IVF will receive everything in the investigator's current ERAS protocol except the home intravenous fluid program. Patients without preexisting vascular access will not receive a midline catheter post-operatively, however the participant will still receive home care for skilled nursing who will provide wound care, ostomy teaching, and education about perioperative fluid management.

No other standard pre-, peri- or post-operative urologic surgery procedures will be affected. Routine care includes an initial clinic consultation, physical examination, and informed consent prior to proceeding with surgery. Informed consent for participation in the study may also be obtained in the preoperative area during the day of surgery. Eligibility will be confirmed at the time of consent. Post- operatively, patients will be given the option of returning to the Johns Hopkins clinic or local follow-up for further ostomy teaching and wound check approximately 7-14 days after surgery. Discussions about the surgical specimen's pathology and initiation of potential adjuvant therapy will not be impacted. All patients will receive phone calls at 30 and 90 days post operatively to assess for complications, emergency department visits, and hospital re-admissions using a standardized template.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than 18 years of age and older
* Confirmed urothelial carcinoma on pathology, including muscle invasive, non-muscle invasive, and variant histology
* Patient electing to undergo radical cystectomy with bilateral pelvic lymphadenectomy after counseling with a urologic oncologist.

Exclusion Criteria:

* Patients undergoing radical cystectomy for benign indications (e.g. chronic bladder pain, fistulas, severe lower urinary tract symptoms)
* Patients undergoing radical cystectomy for a non-bladder primary malignancy (e.g. rectal, colon, uterine cancers).
* Patients with extensive locally advanced disease necessitating a pelvic exenteration
* Contraindication to receiving home IVF therapy (i.e. pre-existing cardiac, renal, hepatic dysfunction)
* Unwilling or unable to participate in 30 and 90 day follow-up phone calls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with 90-day Hospital Readmission | From date of surgery up to 90-days postoperatively
  The primary outcome will be 90-day hospital readmissions that are unplanned, including admissions for observation

SECONDARY OUTCOMES:
Percentage of participants with 30-day hospital readmissions | From date of surgery up to 30-days post-operatively
  The percentage of patients with unplanned hospital readmission within 30 days post-discharge after surgery
Percentage of participants with 90-day emergency department presentations | From date of surgery up to 90 days after surgery
  The percentage of patients with presentations to the emergency department within 90 days after surgery
Percentage of participants with All-cause Complications | From surgery up to 90 days post surgery
  All-cause complications including complications related to the surgery like bleeding, infection, Acute Kidney Injury (AKI), failure to thrive, and complications related to midline or port venous access including infection and thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Max Kates, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No